CLINICAL TRIAL: NCT00905593
Title: An Open-label, Multicenter Study Providing Continuation of Nilotinib in Adult Patients With Imatinib-(Glivec®/Gleevec®) - Resistant or - Intolerant Chronic Myeloid Leukemia in Blast Crisis, Accelerated Phase or Chronic Phase
Brief Title: Nilotinib in Adult Patients With Imatinib-resistant or Intolerant Chronic Myeloid Leukemia in Blast Crisis, Accelerated Phase or Chronic Phase
Acronym: ENACT
Status: Approved for marketing | Type: Expanded Access
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAMN107AMX01
Record Dates: First submitted 2009-05-18; First posted 2009-05-20 (Estimated); Last update posted 2012-07-18 (Estimated); Status verified 2012-07

CONDITIONS: Chronic Myeloid Leukemia
Keywords: chronic myeloid leukemia,; blast crisis,; accelerated phase,; nilotinib,; imatinib,; resistant,; intolerant,; chronic phase
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Blast Crisis | interventions — nilotinib

INTERVENTIONS:
Drug: Nilotinib

SUMMARY:
Multi-center, open-label, non-randomized trial to evaluate long-term safety and efficacy of nilotinib. Approximately 20 patients will be enrolled in this trial at 3 centers in Mexico, which means all ongoing patients participating on [CAMN107A2109] excluding discontinued patients. During this study, patients will receive nilotinib orally, at a dose of 400 mg b.i.d. Patients will normally receive nilotinib on an outpatient basis. This trial will have a maximum of 24 months of follow-up time.

ELIGIBILITY:
Inclusion Criteria:

* Having participated in Novartis study CAMN107A2109, and
* Written signed and dated informed consent prior to any study procedures being performed.

Exclusion Criteria:

* Impaired cardiac function,
* Use of therapeutic coumarin derivatives (i.e., warfarin, acenocoumarol, phenprocoumon) up to the day before study drug administration; Other concurrent severe and/or uncontrolled medical conditions,
* Patients who are currently receiving treatment with any of the medications that have the potential to prolong the QT interval,
* patients who have undergone a major surgery and have not recovered from side effects of such therapy within 15 days,
* Patients who are pregnant or breast feeding or adults of reproductive potential not employing an effective method of birth control, OR
* Patients unwilling or unable to comply with the protocol.

Other protocol -defined inclusion/exclusion criteria may apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 2008-09; Primary Completion 2011-04 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (2):
- Mexico (2):
  - Novartis Investigative Site, Guadalajara, Jalisco
  - Novartis Investigative Site, Mexico City